CLINICAL TRIAL: NCT07394387
Title: A Single-Center, Phase II Clinical Study of HIFU With or Without PD-1 Inhibitors Followed by Abraxane Plus Carboplatin Neoadjuvant Therapy in Triple-Negative Breast Cancer.
Brief Title: Neoadjuvant Study of HIFU With or Without PD-1 Inhibitors Followed by Abraxane Plus Carboplatin in Triple-Negative Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJMU-BC05
Record Dates: First submitted 2025-11-24; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sintilimab; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a single-center, phase II study with two parallel, non-randomized cohorts. Participants are assigned to one of the following intervention sequences based on investigator discretion and clinical considerations:
  Cohort A: Receives High-Intensity Focused Ultrasound (HIFU) sparse scanning. Two weeks later, they begin 6 cycles of neoadjuvant therapy with albumin-bound paclitaxel + carboplatin + the PD-1 inhibitor Sintilimab.
  Cohort B: Receives High-Intensity Focused Ultrasound (HIFU) sparse scanning combined with a single dose of the PD-1 inhibitor Sintilimab. Two weeks later, they begin 6 cycles of neoadjuvant therapy with albumin-bound paclitaxel + carboplatin + Sintilimab.
  The primary distinction between the cohorts is the timing of the first dose of Sintilimab (before vs. concurrent with chemotherapy).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (HIFU + Chemo + PD-1 Inhibitor) (Experimental)
  Interventions: Drug: Sintilimab; Drug: Abraxane; Drug: Carboplatin; Procedure: High-intensity focused ultrasound (HIFU)
- Cohort B (HIFU + PD-1 Inhibitor → Chemo + PD-1 Inhibitor) (Experimental)
  Interventions: Drug: Sintilimab; Drug: Abraxane; Drug: Carboplatin; Procedure: High-intensity focused ultrasound (HIFU)

INTERVENTIONS:
Drug: Sintilimab — 200 mg, administered intravenously every 3 weeks.
Drug: Abraxane — 260 mg/m², administered intravenously on Day 1 of each 21-day cycle.
Drug: Carboplatin — AUC = 6, administered intravenously on Day 1 of each 21-day cycle.
Procedure: High-intensity focused ultrasound (HIFU) — HIFU sparse scanning. Under ultrasound guidance, the tumor and a 5mm margin of surrounding normal tissue are ablated using a point-by-point protocol (150W power, 3s irradiation per point, 5mm point spacing). Performed once.

SUMMARY:
Background:

Triple-negative breast cancer (TNBC) is an aggressive type of breast cancer with limited treatment options. Research suggests that using High-Intensity Focused Ultrasound (HIFU) to destroy the tumor and/or PD-1 inhibitor drugs to activate the immune system before starting chemotherapy may improve treatment effectiveness. This study aims to investigate this new approach.

Objective:

To evaluate the effectiveness and safety of using HIFU, with or without a PD-1 inhibitor (Sintilimab), before and during combination chemotherapy in patients with early-stage TNBC. The primary goal is to determine if this strategy can increase the rate of pathological complete response (pCR).

Study Design:

This is a single-center, Phase II clinical study. Approximately 40 participants with Stage II-III TNBC will be enrolled and assigned to one of two groups (cohorts) without randomization:

Cohort A: Receives HIFU treatment. Two weeks later, begins standard chemotherapy (Abraxane and carboplatin) combined with the PD-1 inhibitor Sintilimab for 6 cycles.

Cohort B: Receives HIFU treatment combined with a single dose of the PD-1 inhibitor Sintilimab. Two weeks later, begins the same 6 cycles of chemotherapy (Abraxane and carboplatin) combined with Sintilimab.

Main Measures:

The primary measure is the rate of pathological complete response (pCR), defined as the absence of invasive cancer in the breast and lymph nodes after surgery following the completion of neoadjuvant therapy.

Other important measures include:

The ability of the treatment to activate the immune system (measured by changes in CD8+ T cells or IFN-γ).

The percentage of patients whose tumors shrink significantly (Objective Response Rate).

How long patients live without their cancer getting worse (Event-Free Survival).

The rate of patients who can undergo breast-conserving surgery. The frequency and severity of side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 and ≤65 years.
2. Histologically confirmed invasive breast cancer, classified as Stage II-III triple-negative breast cancer (TNBC) according to the 8th edition AJCC TNM staging.
3. At least one measurable lesion as per RECIST v1.1 criteria.
4. No prior chemotherapy, immunotherapy, endocrine therapy, radical surgery, or radiotherapy for breast cancer.
5. ECOG performance status of 0 or 1.
6. Adequate organ function, defined as:

   * Hemoglobin ≥90 g/L
   * White blood cell count ≥3.5×10^9/L
   * Platelet count ≥100×10^9/L
   * Absolute neutrophil count ≥1.5×10^9/L
   * AST and ALT ≤3× upper limit of normal (ULN)
   * Total bilirubin ≤1.5× ULN
   * Serum creatinine ≤1.5× ULN
   * No evidence of pneumonia on chest CT
7. Adequate cardiac function, defined as:

   * No myocardial ischemia on ECG
   * NYHA class I
   * LVEF ≥55% on echocardiogram
   * Normal cardiac markers (cTnI and BNP)
8. Normal thyroid function (T3, T4, FT3, FT4, TSH).
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Male or inflammatory breast cancer.
2. Metastatic (Stage IV) breast cancer.
3. History of active autoimmune or inflammatory diseases requiring systemic treatment within the past 2 years (e.g., systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis). Exceptions: type I diabetes, hypothyroidism controlled with hormone replacement therapy, or skin disorders not requiring systemic treatment (e.g., vitiligo, psoriasis).
4. Concurrent other malignancies or history of other malignancies within the past 5 years (except adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix).
5. Any other serious non-malignant disease that may compromise compliance or place the patient at risk.
6. Major surgery within 4 weeks prior to study initiation or anticipated need for major surgery during the study.
7. Prior radiotherapy, chemotherapy, targeted therapy, endocrine therapy, or major surgery for breast cancer.
8. Known hypersensitivity to any component of the study drugs.
9. Poorly controlled cardiac disease (e.g., NYHA class II+ heart failure, unstable angina, myocardial infarction within the past year, or clinically significant arrhythmias requiring intervention).
10. History of interstitial lung disease (ILD), current ILD, or suspected ILD on imaging during screening.
11. Active infections, including:

    * HIV positive
    * Active tuberculosis
    * Active hepatitis B (HBV-DNA > 10^3 IU/mL)
    * Active hepatitis C (HCV antibody positive with detectable HCV-RNA)
12. Active autoimmune disease requiring systemic treatment.
13. Dementia, significant intellectual impairment, or any psychiatric condition that impairs understanding of the informed consent.
14. Unhealed wounds, ulcers, or fractures within 4 weeks prior to signing consent; or any history of clinically significant bleeding or bleeding tendency.
15. Any other condition deemed by the investigator to be unsuitable for trial participation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Proportion of participants with a ≥2-fold increase in CD8+ T cell count or IFN-γ level | 2 weeks after HIFU treatment (and concurrent PD-1 inhibitor for Cohort B), which is immediately prior to the start of the first cycle of neoadjuvant chemotherapy.
Objective Response Rate (ORR) | Every 6 weeks during neoadjuvant therapy (at the end of cycles 2, 4, 6), up to up to 24 weeks
Event-Free Survival (EFS) | From enrollment until the first occurrence of an event, assessed up to 5 years.
Breast-Conserving Surgery (BCS) Rate | through study completion, an average of 1 year
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline, 1 month post-intervention, 6 months post-intervention and at study completion (an average of 1 year)

OTHER OUTCOMES:
Overall Survival (OS) | From enrollment until death, assessed up to 5 years.
predictive biomarkers for treatment efficacy | Biomarker samples are collected at baseline (pre-treatment) and at surgery (post-neoadjuvant therapy). Analysis will be performed after completion of patient enrollment and follow-up, through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Bianchini G, De Angelis C, Licata L, Gianni L. Treatment landscape of triple-negative breast cancer - expanded options, evolving needs. Nat Rev Clin Oncol. 2022 Feb;19(2):91-113. doi: 10.1038/s41571-021-00565-2. Epub 2021 Nov 9. PMID 34754128
- [Background] Hu Z, Yang XY, Liu Y, Morse MA, Lyerly HK, Clay TM, Zhong P. Release of endogenous danger signals from HIFU-treated tumor cells and their stimulatory effects on APCs. Biochem Biophys Res Commun. 2005 Sep 16;335(1):124-31. doi: 10.1016/j.bbrc.2005.07.071. PMID 16055092
- [Background] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663